CLINICAL TRIAL: NCT06200181
Title: Effect of Olanzapine on Opioid Craving and Misuse Among Patients Receiving Opioids for Cancer-related Pain: A Pilot Double-Blind, Randomized Control Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-0492; NCI-2023-11092 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Misuse, Opioid
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1 (Experimental): Participants will take a lower dose of olanzapine every day for Days 1-7 and then a higher dose every day for the next 3 weeks
  Interventions: Drug: Olanzapine
- Arm 2 (Experimental): Participants will take the lower dose of olanzapine every day for 4 weeks.
  Interventions: Drug: Olanzapine
- Arm 3 (Placebo Comparator): Participants will take a placebo every day for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olanzapine — Given by PO
  Other Names: Zypreza
  Arms: Arm 1
Drug: Olanzapine — Given by PO
  Other Names: Zypreza
  Arms: Arm 2
Drug: Placebo — Given by PO
  Arms: Arm 3

SUMMARY:
To learn about the effectiveness of taking the antipsychotic medication olanzapine to help lower opioid craving.

DETAILED DESCRIPTION:
Primary Objective To determine the effect of olanzapine on opioid craving among patients receiving opioids for cancer pain (Opioid Craving Scale; Opioid Craving Visual Analogue Scale, change from baseline)

Secondary Objective To determine the effect of olanzapine on opioid misuse among patients receiving opioids for cancer pain (Current Opioid Misuse Measure, change from baseline)

Exploratory Objective

* To estimate the effect of olanzapine and placebo on the amount of opioid use among patients receiving opioids for cancer pain (morphine equivalent daily dose)
* To determine the effect of olanzapine and placebo on pain intensity among patients receiving opioids for cancer pain (Brief Pain Inventory)
* To determine the effect of olanzapine and placebo on overall symptom burden among patients receiving opioids for cancer pain (ESAS symptom Distress Score)
* To estimate the differences between the olanzapine and placebo effects on opioid craving and misuse measures (Opioid Craving Scale, Opioid Craving Visual Analogue Scale, Current Opioid Misuse Measure)
* To determine the adverse effects of olanzapine and placebo among patients receiving opioids for cancer pain (National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0)

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Diagnosis of cancer pain
3. Receiving long-term opioid therapy (≥ 7 days)32
4. Active use of opioids within the past 7 days
5. Opioid misuse behavior (COMM score ≥ 9/68)
6. Seen by a Supportive Care Clinic or Pain Clinic clinician
7. ECOG performance status ≥ 2/4
8. Ability to communicate in English
9. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Contraindications to, or allergic to, olanzapine
2. Current use of any antipsychotic medication (e.g. quetiapine, haloperidol, risperidone, etc.)
3. History of OUD or other substance use disorders, except marijuana
4. History of formal psychiatric diagnoses (e.g. bipolar disorder, schizophrenia, major depressive disorder, or anorexia nervosa)
5. Hepatic insufficiency (defined as alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 times the highest normal value, or total bilirubin >1.5 times the highest normal value) within the past month
6. History of uncontrolled Diabetes Mellitus or hyperglycemia (fasting ≥ 200 mg/dL) within the past month
7. History of seizure disorder or neuroleptic malignant syndrome
8. History of cardiac disease (e.g. coronary artery disease, congestive heart failure)
9. (Females only) Known pregnancy, as communicated to study personnel by clinicians; females of childbearing potential will receive advice to use methods of contraception per usual care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Arthur, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org